CLINICAL TRIAL: NCT07031258
Title: Prospective Real-world Data Evaluation of Darolutamide (DARO) in Combination With Androgen-deprivation Therapy (ADT) and Docetaxel (DOC) in Patients With Metastatic Hormone-sensitive Prostate Cancer
Brief Title: Evaluation of the Efficacy of Darolutamide Triplet Therapy in Patients With Metastatic Hormone-sensitive Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-218
Record Dates: First submitted 2025-05-28; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer; Darolutamide (DARO) in Combination With Androgen-deprivation Therapy (ADT) and Docetaxel (DOC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dose of docetaxel — According to the relative dose intensity of docetaxel (RDI; Defined as the ratio of the dose received to the full planned dose of 75mg/m2 per 6 cycles specified in the protocol) were divided into cohort 1 (patients receiving docetaxel dose intensity ≤80%) and cohort 2 (patients receiving docetaxel dose intensity ≤80%). A total of 50 patients who received docetaxel dose intensity > 80% were planned to be enrolled, including 25 patients in the docetaxel dose intensity ≤80% group and 25 patients in the docetaxel dose intensity > 80% group

SUMMARY:
The purpose of this study is to investigate the clinical efficacy and safety of darolutamide combined with androgen deprivation therapy (ADT) and different dose-intensity docetaxel chemotherapy in the treatment of patients with metastatic hormone-sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily signed informed consent form and able to understand and agree to comply with study requirements; Age ≥18； Male； Patients diagnosed with metastatic hormone-sensitive prostate cancer via CSCO guidelines, histopathology, etc.； Patients determined by treating physician to require darolutamide triplet therapy ECOG performance status score of 0-1 as evaluated by the Eastern Cooperative Oncology Group (ECOG) criteria； Life expectancy of over 1 year； Good compliance with regular serum PSA testing during treatment；

Exclusion Criteria:

Presence of other malignancies within the past 2 years or currently; Severe cardiovascular/cerebrovascular disease within 6 months prior to study treatment initiation, including: severe/unstable angina, myocardial infarction, congestive heart failure [NYHA Class III or worse], stroke, or arrhythmia requiring medication; Allergy to any study drug or excipient; Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors affecting drug intake/absorption; Underlying medical condition/alcohol or drug abuse/dependence that may interfere with drug administration, result in adverse events, or complicate outcome interpretation; Participation in another therapeutic clinical study; Deemed unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with metastatic hormone-sensitive prostate cancer who have chosen to receive darolutamide triplet therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
6-month prostate-specific antigen (PSA) undetectable rate | From the beginning of the patient's treatment to 6 months
  The proportion of patients with PSA <0.2 ng/mL after 6 months of treatment

SECONDARY OUTCOMES:
Radiological progression-free survival | From the beginning of the patient's treatment to 6 months
  Time from treatment initiation to radiological progression
PSA kinetics curve | Every 3 weeks during the triplet therapy, and every month after treatment.
  The PSA decline curve from the start of ADT, darolutamide, and docetaxel treatment to the completion of docetaxel.

IPD SHARING:
Plan to Share IPD: No